CLINICAL TRIAL: NCT07132073
Title: MR-guided Brachytherapy and SBRT for Unfavorable Prostate Cancer
Brief Title: MRI-guided Locoregional SBRT Prostate Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024.199
Record Dates: First submitted 2025-08-12; First posted 2025-08-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: SBRT; brachytherapy; MR-guided irradiation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation Phase (Experimental): Brachytherapy + MR-guided SBRT
  Interventions: Radiation: Brachytherapy + SBRT

INTERVENTIONS:
Radiation: Brachytherapy + SBRT — Brachytherapy + SBRT

SUMMARY:
The implementation of Magnetic Resonance Image Guided Radiotherapy (MRgRT) into a Prostate Cancer Program will allow to reproduce the results obtained with state-of-the-art brachytherapy combined with EBRT with the added advantage of convenience.

DETAILED DESCRIPTION:
The implementation of Magnetic Resonance Image Guided Radiotherapy (MRgRT) into a Prostate Cancer Program will allow to reproduce the results obtained with state-of-the-art brachytherapy combined with EBRT with the added advantage of convenience.

Rationale In the radiation setting, MRI provides superior soft tissue contrast compared to standard onboard X-ray imaging improving inter- and intra- observer delineation variation. MRgRT offers the opportunity to adapt the plan at each fraction to the anatomical changes seen. This is especially important in prostate cancer where the prostate is subject to large intra and/or interfractional position changes due to rectal and bladder filling changes.

Primary Objectives A. To achieve a 5-year biochemical relapse-free survival of 85%. B. To decrease urinary grade 3 or greater toxicity below 5% and rectal grade 3 or greater toxicity below 2%.

Secondary Objectives A. Determination of blood and urine biomarkers of treatment response and toxicity .

B. Determination of radiomics biomarkers of treatment response and toxicity . C. Determination of QOL with IPSS and EORTC QLQ-PR25

ELIGIBILITY:
Inclusion Criteria:

* Patients with unfavorable intermediate, high and very high risk PCa as per the NCCN stratification criteria .
* Suboptimal candidates for high-dose therapy such as elderly, frail patients or patients with large volume glands (i.e, >60cm3) or extensive TURP in the prior 6-12 months should be considered cautionary indications.
* Patients with low risk of nodal spread may be treated on a MRI-guided local SBRT program.

Exclusion Criteria:

* No prior radiation therapy to the target areas
* Patient able to undergo a MRI exam

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical relapse-free survival | 5-years
  To achieve a 5-year biochemical relapse-free survival of 85%.

SECONDARY OUTCOMES:
Adverse Events | 5-years
  To decrease urinary grade 3 or greater toxicity below 5% and rectal grade 3 or greater toxicity below 2%.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Martínez-Monge, M.D., Principal Investigator — Clínica Universidad de Navarra; Luis Fuertes, M.D., Principal Investigator — Clínica Universidad de Navarra

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5-years
Access Criteria: On request